CLINICAL TRIAL: NCT04691466
Title: Assessment of Clinical Outcome Following Total Hip and Knee Replacement
Brief Title: Study Evaluating the Efficacy of Joint Replacement
Acronym: SEVERE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicolaus Copernicus University (Other)
Collaborators: Warmia and Mazury Oncology Centre (Unknown)
Responsible Party: Principal Investigator, Przemyslaw Paradowski, M.D., Ph.D., Nicolaus Copernicus University
Other Study IDs: WN758
Record Dates: First submitted 2020-12-27; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Replacement; Arthroplasty; Patient-relevant outcome measure (PROM); KOOS; HOOS
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Arthroplasty, Replacement; Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIP_R: Patients undergoing hip replacement surgery
  Interventions: Procedure: Joint replacement
- KNEE_R: Patients undergoing knee replacement surgery
  Interventions: Procedure: Joint replacement

INTERVENTIONS:
Procedure: Joint replacement — Routinely performed hip- or knee replacement
  Other Names: Joint arthroplasty

SUMMARY:
Patient-related outcomes were originally designed to measure outcomes in clinical studies. They were not developed to predict outcomes, however, different studies showed close association between values achieved preoperatively and postoperative outcomes. The aim of the present trial is to identify patients with satisfactory and unsatisfactory outcomes after joint replacement and to investigate whether there are any potential predicting potential in preoperative results of the patient-related outcomes and if there exist other predicting factors for functional recovery or treatment failure after joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients with primary or secondary hip- and knee osteoarthritis undergoing joint replacement surgery.

Exclusion Criteria:

1. An inability to understand the Polish language,
2. Presence of neuromuscular disease and cognitive impairment,
3. Having a prosthesis in another joint of the ipsilateral or contralateral lower limb placed within 6 months before the current surgery,
4. Having rheumatoid arthritis,
5. Symptoms in several joints (hip, knee or ankle) with expected total joint arthroplasty within 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with osteoarthritis of the hip or knee.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the patients' opinion about their hip. Change over time | 12 months
  Change between the following assessments as measured with the Hip disability and Osteoarthritis Outcome Score (HOOS) in patients undergoing total hip replacement; 0-100 points, worst to best; minimal clinical difference (MCD) = 10 points.
Assessment of the patients' opinion about their knee. Score change over time | 12 months
  Change between the following assessments as measured with the Knee injury and Osteoarthritis Outcome Score (KOOS) in patients undergoing total knee replacement; 0-100 points, worst to best; minimal clinical difference (MCD) = 10 points.

SECONDARY OUTCOMES:
Assessment of the quality of life. Score change over time | 12 months
  Results of the generic PROM, the Short Form Health Survey-36 (SF-36) in both, patients undergoing hip and knee replacement; 0-100 points, worst to best.
Pain intensity. Change over time | 12 months
  Measured with the Visual Analog Scale (VAS); 0-10 points, worst to best.
Hip abductors muscle strength. Change over time | 12 months
  Determination of the Trendelenburg's sign in patients undergoing total hip replacement in following assessments; positive or negative.
Range of motion. | 12 months
  Assessment of range of motion in hips and knees, respectively, in following assessments; degrees.

OTHER OUTCOMES:
Body mass index (BMI) | 12 months
  Measurement of weight in kilograms and height in meters to combined to report BMI in kg/m^2; to be measured twice, before intervention and after 12 months.
Activity | 12 months
  Measured with the Tegner Activity Score (TAS); 1-10 points, worst to best; to be measured twice, before intervention and after 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwik Rydygier Collegium Medicum, Faculty of Health Sciences, Jagiellońska 13/15, Bydgoszcz, Poland